CLINICAL TRIAL: NCT00314301
Title: Motion Analysis of Sit-to-Stand Movements in Children With Spastic Diplegia Before and After Loaded Sit-to-Stand Training
Brief Title: Motion Analysis of Sit-to-Stand Movements in Children With Spastic Diplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 94023
Record Dates: First submitted 2006-04-12; First posted 2006-04-13 (Estimated); Last update posted 2006-04-17 (Estimated); Status verified 2006-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; resistance; movement; biomechanics
MeSH Terms: conditions — Cerebral Palsy

INTERVENTIONS:
Device: loaded sit-to-stand training

SUMMARY:
The purpose of this study is to compare movement variations before and after the loaded training, with kinematics, kinetics, and electromyography, in children with spastic diplegia and to further discuss mechanisms of the loaded training.

DETAILED DESCRIPTION:
Subjects: This study will recruit twenty children who are aged between 5 and 12 years, with spastic diplegia, and without having major surgeries or botulinum toxin injection on lower extremities during the past 6 months prior to participate in this study.

Methods: The Vicon 250 motion analysis system, 3 AMTI force platforms and the EMG recording system will be used to collect data of sit-to-stand (STS) movements. Baseline, pre- and post-training evaluations will be carried out. The duration of the baseline and pre-training evaluations is 2 months. The training period will take about 6 weeks. Each evaluation will take two separate days to accomplish. On the first day, the STS1RM of individual children was determined. On the second day, kinematic and kinetic data of STS movements in natural and loaded (applying load of 50% STS1RM during STS movements) conditions were collected. Data of smoothness, maximal extension moment and around hip and knee joints, onset time of lower extremity muscles will then be calculated. Results of each evaluation will be used for further comparison.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as spastic diplegia
* Aged between 5 and 12 years
* Able to perform the STS movements without assistance
* Able to cooperate and understand commands given

Exclusion Criteria:

* Severe musculoskeletal deformity or pain on lower extremities
* Botulism injection in the past 3 months or major operations in the preceding 6 months on lower extremities
* Uncontrolled epilepsy
* Major sensory deficits, such as blindness or deafness

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2006-04; Study Completion 2007-09

PRIMARY OUTCOMES:
kinematic measures of lower extremity and the whole body
kinetic measures of lower extremity and the whole body
electromyographic measures of lower extremity and the whole body

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Ting Lin, MSc, Principal Investigator — Research Ethics Review Committee of the Far Eastern Memorial Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan